CLINICAL TRIAL: NCT02558413
Title: A Double-Blind, Placebo-Controlled, Single Ascending Oral Dose Study of the Safety and Pharmacokinetics of BTA-C585 in Healthy Volunteers
Brief Title: Phase 1 Safety and Pharmacokinetics Study of Single Ascending Doses of BTA-C585 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biota Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Vaxart (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTA585-001
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Pharmacokinetics; Healthy Volunteers
Keywords: Viral Diseases; Antiviral; Paramyxoviridae Infections; RSV; Respiratory Syncytial Virus; Aviragen Therapeutics, Inc.; Aviragen Therapeutics; Aviragen
MeSH Terms: conditions — Virus Diseases; Paramyxoviridae Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BTA-C585 oral capsules (Active Comparator): 25 or 100 mg oral capsules; Single ascending doses (SAD) from 50 mg to 800 mg
  Interventions: Drug: BTA-C585 oral capsules
- BTA-C585 matching placebo (Placebo Comparator): BTA-C585 Matching placebo capsules; single doses
  Interventions: Drug: BTA-C585 matching placebo

INTERVENTIONS:
Drug: BTA-C585 oral capsules — BTA-C585; Single ascending doses from 50 mg to 800 mg
  Other Names: BTA585
  Arms: BTA-C585 oral capsules
Drug: BTA-C585 matching placebo — Single ascending doses to match 50 to 800 mg BTA-C585 capsules
  Other Names: BTA585
  Arms: BTA-C585 matching placebo

SUMMARY:
This is a placebo-controlled, double-blind, randomized, single dose escalation Phase 1 clinical trial to determine the safety and tolerability of BTA-C585 administered orally to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged 18-60 years;
* Weight ≥ 50 kg and Body Mass Index (BMI) of 19 to 32;
* Female subjects must be of non-childbearing potential;
* Male subjects must agree to use a double barrier method of birth control;
* Able to provide informed consent

Exclusion Criteria:

* Current or recent (within 14 days of Day 0) bacterial or viral infection;
* Positive results for hepatitis B, hepatitis C, or HIV;
* Clinically significant abnormalities noted on ECG;
* Safety laboratory abnormalities;
* Regular use of medications, prescription or non-prescription;
* Poor vein access or fear of venipuncture;
* Major surgery, significant recent injury or trauma within 30 days;
* Received an investigational drug or vaccine within 30 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | Day 0 to Day 11
Area under the plasma concentration-time curve (AUC) from time 0 to 24 hours | 0-24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Anna Novotney-Barry, Study Director — Biota Pharmaceuticals, Inc.
Locations (1):
- Biota Investigational Site, San Antonio, Texas, United States